CLINICAL TRIAL: NCT04377373
Title: Correlation Between Sacral Angle and Lumbar Range of Motion in Women With Genu Valgum
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima Abdelaty Hassan, Lecturer, Cairo University
Other Study IDs: P.T.REC/012/002300
Record Dates: First submitted 2019-09-06; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Genu Valgum
MeSH Terms: conditions — Genu Valgum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many patients with genu valgum present with postural changes, such as: internal rotation of the tibial and femoral axes, anteversion of the iliac bones, increased lumbar lordosis, thoracic hyperkyphosis and cervical hyperlordosis. Such pathomechanical changes may interfere with lumbar range of motion. Investigators of this study try to answer the following question: is there a relationship between sacral angle and lumbar range of motion in women with bilateral genu valgum. the results of this study will help professionals to plan a proper treatment program for patients with genu valgum.

DETAILED DESCRIPTION:
Sixty four female participants were under the following procedures:

* Screening for genu valgum via postural assessment from frontal view, then measuring the Q angle bilaterally.
* Patients with Q-angle >20 degress were under the following procedures:

A. Full-Length AP standing X-ray,then the investigators measured the hip-knee angle (the angle between the mechanical axis of the femur and the tibia). It will be obtained by connecting the center of the femoral head to the midpoint of the tibial eminential spine in a line tangential to the femoral condyles, and another line from here to the centre of the trochlea tali.

B-Lumbo-sacral X-ray lateral view was done at the time and the sacral angle was the measured by Ferguson´s technique in degrees using a protractor and this was the sacral angle.

C- During the same session, trunk range of motion was measured by Modified schober test D- Collected data were taken for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Female with bilateral genu valgum (Q angle> 20 degrees.
2. Age ranges from 18-25 years old.
3. BMI ≥ 30 (kg/m2)

Exclusion Criteria:

1. Previous lumbar surgery
2. lumbar spine fracture
3. Spondylolisthesis
4. Foraminal or extra foraminal lumbar disc herniation
5. spinal tumors, and bone metabolic diseases 6 - Knee surgeries

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female with bilateral genu valgum with age range 18-25 and BMI≥ 30 (kg/m2)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Sacral angle | 30 minutes
  After X-ray lateral view for lumbo-sacral spine, the investigators used a 30 cm long transparent ruler to measure the sacral angle on the X-ray film.
  Two lines were drawn, the first line along the superior margin of the sacrum, and the second line was the horizontal line.
  The acute angle between 2 lines(sacral angle) was measured in degrees using a protractor.
Lumbar range of motion measured by Modified Shobber test | 15 minutes
  * Patient was directed to stand with the back exposed.
  * Dimples of Venus (posterior superior iliac spine) was determined and was marked by pertinent marker.
  * Using tape measurement, the researcher marked a point 5 cm below and 10 cm above marked dimples (total marked area was 15 cm).
  * Then the subject was asked to lean forward without bending the knees.
  * The distance between 2 points was measured (D), then the ROM was determined by the following equation; ROM = D -15.

CONTACTS AND LOCATIONS:
Overall Officials: Nasr A. Abdelkader, PhD, Principal Investigator — Lecturer,Cairo University
Locations (1):
- Cairo university, Giza, Egypt